CLINICAL TRIAL: NCT06744569
Title: A Randomized, Double-blind, Vehicle-Controlled Phase I Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetic Profile and Preliminary Efficacy of CU-10101 Unguent in Healthy and AD Participants
Brief Title: A Phase I Clinical Trial to Evaluate CU-10101 Unguent
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Cutia Therapeutics（Wuxi）Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CU-10101-103
Record Dates: First submitted 2024-08-09; First posted 2024-12-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Atopic Dermatitis
Keywords: CU-10101 unguent
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Part1: cohort1 (Experimental): BSA20%_0.3% (10g:30mg)
  Interventions: Drug: CU-10101
- Part1: cohort2 (Experimental): BSA20%_1%(10g:100mg)
  Interventions: Drug: CU-10101
- Part1: cohort3 (Experimental): BSA20%_2%(10g:200mg)
  Interventions: Drug: CU-10101
- Part1: cohort4 (Experimental): BSA40%_2%(10g:200mg)
  Interventions: Drug: CU-10101
- Part2: cohort1 (Experimental): QD_0.3%(10g:30mg)
  Interventions: Drug: CU-10101
- Part2: cohort2 (Experimental): QD_1%(10g:100mg)
  Interventions: Drug: CU-10101
- Part2: cohort3 (Experimental): QD_2%(10g:200mg)
  Interventions: Drug: CU-10101
- Part2: cohort4 (Experimental): BID_2%(10g:200mg) or BID_1%(10g:100mg)
  Interventions: Drug: CU-10101

INTERVENTIONS:
Drug: CU-10101 — 0.3%CU-10101 ；1%CU-10101 ；2%CU-10101； Placebo

SUMMARY:
The study was conducted in two parts:Part 1 and Part 2.Part 1 is a single-site,randomized,double-blind,vehicle-controlled single and multiple administration,dose-escalation study in healthy Chinese participants.There are four cohorts in Part 1.Part 2 is a randomized,double-blind,vehicle-controlled single and multiple administration,dose-escalation study in Chinese participants with mild to moderate atopic dermatitis.It is planned to be conduct in 1 to 3 sites,with a total of four cohorts in Part 2.

DETAILED DESCRIPTION:
Part 1:This is a randomized, double-blind, vehicle-controlled Phase I clinical trial to evaluate the safety, tolerability, and pharmacokinetic profile of CU-10101 unguent after single and multiple doses in adult healthy subjects. The study consisted of screening, dosing, and end-of-study (EOS) visits.

Screening (D-7 to D-1): from 7 days before dosing (D-7) to 1 day prior to dosing (D-1), subjects will undergo screening-related examinations as required by this protocol after signing the informed consent form, and eligibility will be confirmed according to the inclusion/exclusion criteria. Eligible subjects will be admitted to the Phase I clinical trial site 1 day before dosing (D-1), relevant examinations will be performed as required by the protocol, and the inclusion/exclusion criteria will be confirmed again. Reconfirmed eligible subjects will remain in the study. Draw areas of skin that require drug application based on body maps .

Dosing period (D1-D13): Subjects will be randomized prior to dosing on D1 (each cohort will be randomized in a 2: 1 ratio to the investigational product or vehicle group) and CU-10101 unguent or vehicle will be evenly applied to the specified dose position on the morning of D1 and every morning (dosing interval is 24 h ± 0.5 h) from D4 to D10 based on randomization results. Subjects will collect PK blood samples at the time points specified in the protocol. Left the Phase 1 clinical site after completing blood sampling and relevant examinations on D13.

EOS Visit period (D20): Subjects will return to the Phase I clinical trial site for safety monitoring on D20 ± 1.

Part 2

This is a randomized, double-blind, vehicle-controlled Phase 1 clinical trial to evaluate the safety, tolerability, and pharmacokinetic profile of CU-10101 unguent after single and multiple doses in adult subjects with atopic dermatitis meanwhile exploring efficacy after multiple doses. The study consisted of screening, dosing, and end-of-study (EOS) visits.

Screening (D-14 to D-1): from 14 days before dosing (D-14) to 2 days prior to dosing (D-2), subjects will undergo screening-related examinations as required by this protocol after signing the informed consent form, and eligibility will be confirmed according to the inclusion/exclusion criteria. Eligible subjects will be admitted to the Phase I clinical trial site 1 day before dosing (D-1), relevant examinations will be performed as required by the protocol, and the inclusion/exclusion criteria will be confirmed again. Reconfirmed eligible subjects will remain in the study. Draw areas of skin that require drug application based on body maps .

Dosing period (D1-D29): sujects will be randomized prior to dosing on D1 (each cohort will be randomized in a 4: 1 ratio to the investigational product group or vehicle group) and CU-10101 unguent or vehicle will be evenly applied to the skin lesion sites every morning from D1 to D28 based on the randomization results (dosing will be completed by 12：00 noon daily for QD dosing group; dosing will be administered only once on D1 and D7 of BID groups, dosing interval is not less than 8 h). Given that CU-10101 is a high clearance compound, subjects will leave the Phase 1 clinical trial site after completing the single dose to continue multiple doses of CU-10101 unguent or vehicle at the same dose. After complete the relevant examinations and the investigator assesses that the requirements for continuation this trial are met the protocol at the Phase I clinical trial site on D1-D2 and D6-D8, the subjects will continue dosing until the last dose is completed on D28, and the subjects will continue dosing until the study is completed or the treatment discontinuation criteria are met. Subjects returned to the Phase I clinical trial site for safety monitoring and efficacy evaluation on D15 and D29. Safety monitoring included, but was not limited to, vital signs, physical examinations, 12-lead electrocardiograms (ECGs), laboratory examinations (hematology, blood biochemistry, urinalysis), and pregnancy examinations (D29 only), and AEs and concomitant medications. Efficacy evaluations included BSA, IGA score, EASI score, and NRS score. Subjects will collect PK blood samples at the time points. In addition, the skin areas requiring treatment will be redrawn prior to dosing on D8 and D15 and on D29 or the Early Withdrawal Visit.

EOS Visit Period (D36): subjects will return to the Phase I clinical trial site for safety monitoring on D36 ± 1.

ELIGIBILITY:
Inclusion Criteria:

Part 1：1.Subjects were 18-45 years of age (inclusive), male or female, at the time of signing the informed consent form;

2.Male weight ≥ 50.0 kg, female weight ≥ 45.0 kg; body mass index in the range of 18.0-27.0 kg/m2 (including cut-off);

3.Based on physical examination, vital signs, electrocardiogram, and laboratory results, it was shown to be in good health without clinically significant abnormalities (as judged by the investigator);

4.Ability to fully understand the contents of the study, voluntarily participate in the study, and sign the informed consent form. Follow protocol procedures to complete relevant visits during the study;

5.Female participants of childbearing potential and male participants with partners of childbearing potential must consent from signing the informed consent form and no childbearing plan and voluntary use of appropriate contraception up to 3 months after the last dose.

Part 2：1.Subjects were 18-65 years of age (inclusive), male or female, at the time of signing the informed consent form;

2.Diagnosed with AD according to Hanifin-Rajka diagnostic criteria and a history of AD assessed by the investigator for ≥ 6 months;

3.Male weight ≥ 50.0 kg, female weight ≥ 45.0 kg; body mass index in the range of 18.0-27.0 kg/m2 (including cut-off);

4.Investigator Global Assessment (IGA) score of 2 or 3 at screening and baseline;

5.At screening and baseline, BSA was 5% -40% (excluding the area of lesions on the scalp, face, genitalia and intertriginous sites [e.g., axillary, inguinal, elbow fossa, etc.] when calculating the lesion area);

6.Ability to fully understand the contents of the study, voluntarily participate in the study, and sign the informed consent form. Follow protocol procedures to complete relevant visits during the study;

7.Female participants of childbearing potential and male participants with partners of childbearing potential must consent from signing the informed consent form and no childbearing plan and voluntary use of appropriate contraception up to 3 months after the last dose.

Exclusion Criteria:

Part 1 ：1.Allergic constitution (e.g., allergy to two or more drugs, food and pollen), or allergy to the ingredients or excipients of the investigational medicinal product;

2.Those who cannot tolerate venipuncture, or have a history of needle sickness and blood sickness;

3.Subjects with skin damage, atopic dermatitis, eczema, rash, pigmentation and tattoos at the administration site, or other conditions judged by the investigator to be likely to affect drug absorption or affect skin tolerance;

4.Previous or current significant or clinically significant diseases/abnormalities, including, but not limited to, heart/cardiocerebrovascular, respiratory, endocrine, gastrointestinal, kidney, liver, gallbladder, dermatological, hematological, immune, neurological or psychiatric diseases/abnormalities, or, as judged by the investigator, there is a safety risk or impact on safety, tolerability or pharmacokinetic assessment;

5.Participants with a prior diagnosis of malignancy;

6.Lactating women or women with positive pregnancy results, or women who plan to become pregnant during the study;

7.Hepatitis C virus (HCV) antibody, hepatitis B surface antigen (HBsAg), treponema pallidum (TP) antibody, human immunodeficiency virus (HIV) antibody were positive;

8.Those who smoke more than 5 cigarettes per day for 3 months prior to screening or cannot stop using any tobacco products during the study;

9.Frequent drinkers within 3 months prior to screening, i.e., more than 14 units of alcohol per week (1 unit = 360 mL beer or 45 mL of spirits with 40% alcohol or 150 mL of wine) or who were unable to discontinue use of any alcoholic product during the study or had a positive alcohol breath test at screening;

10.Previous history of drug abuse, drug use within 3 months prior to screening, or positive urine drug screen at screening;

11.Donation of blood or massive blood loss (≥ 400 mL) within 3 months prior to screening;

12.Participation in other clinical trials within 3 months prior to screening or during the study;

13.Major surgery within 3 months prior to screening (major surgery is defined in accordance with the Medical Journal of Medicine, May 1, 2009 Grade 3 and 4 surgery specified in the Measures for the Administration of Clinical Application of Therapeutic Techniques), or who plan to undergo surgery during the study;

14.Those who have received live (attenuated) vaccines within 4 weeks prior to screening, or plan to receive live (attenuated) vaccines during treatment and within 4 weeks after the last dose of investigational product;

15.Received any other medication, including herbal and dietary supplements, within 2 weeks or 5 times the elimination half-life prior to screening, whichever is longer;

16.Consumption of excessive amounts of tea, coffee, and/or caffeinated beverages (more than 8 cups, 1 cup = 250 mL) per day for 2 weeks prior to screening;

17.Participants who have taken food or beverages (e.g. grapefruit, grapefruit juice, etc.) or any food or drink containing or metabolized to produce caffeine or xanthine (e.g. coffee, tea, chocolate) within 48 hours prior to dosing;

18.Those who have special requirements for diet and cannot comply with the unified diet;

19.Other conditions or treatments that, as assessed by the investigator, may affect the results of the study, interfere with the participation of participants in the trial, etc.

Part 2：

1. History of allergy to the ingredients or excipients of the investigational product;
2. Those who cannot tolerate venipuncture, or have a history of needle sickness and blood sickness;
3. Previous history of clinically significant cardiac, hepatic, neurological, respiratory, blood, digestive, immune, renal or psychiatric disorders, which, in the opinion of the investigator, increases safety risks, affects safety, tolerability, or pharmacokinetics;
4. Participants with a prior diagnosis of malignancy;
5. Any active skin diseases, such as psoriasis, lupus erythematosus, seborrheic dermatitis, that may have affected the evaluation of the study results;
6. Participants with acute-phase atopic dermatitis whose rash was predominantly erosive, exudative, or had a new skin rash 2 weeks before screening;
7. Active infection or any viral, bacterial, fungal infection (e.g., herpes simplex, herpes zoster, varicella) requiring treatment at screening;
8. Skin lesions were limited to the head, hands, feet, genitalia and intertriginous areas;
9. Lactating women or women with positive pregnancy results, or women who plan to become pregnant during the study;
10. Those who are judged by the investigator to be abnormal and clinically significant at screening or baseline clinical or laboratory tests;
11. Hepatitis C virus (HCV) antibody, hepatitis B surface antigen (HBsAg), treponema pallidum (TP) antibody, human immunodeficiency virus (HIV) antibody were positive;
12. Those who smoke more than 5 cigarettes per day for 3 months prior to screening or cannot stop using any tobacco products during the study;
13. Frequent drinkers within 3 months prior to screening, i.e., more than 14 units of alcohol per week (1 unit = 360 mL beer or 45 mL of spirits with 40% alcohol or 150 mL of wine) or who were unable to discontinue use of any alcoholic product during the study or had a positive alcohol breath test at screening;
14. Previous history of drug abuse, drug use within 3 months prior to screening, or positive urine drug screen at screening;
15. Donation of blood or massive blood loss (≥ 400 mL) within 3 months prior to screening;
16. Participation in other clinical trials within 3 months prior to screening or during the study;
17. Major surgery within 3 months prior to screening (major surgery defined by reference to 01 May 2009 Grade 3 and 4 surgery specified in the Measures for the Administration of Clinical Application of Medical Technology), or who plan to undergo surgery during the study;
18. Those who have received live (attenuated) vaccines within 4 weeks prior to screening, or plan to receive live (attenuated) vaccines during treatment and within 4 weeks after the last dose of investigational product;
19. Systemic systemic therapy (e.g., biologics, small molecule targeted, immunosuppressants, and other systemic therapies, etc.) for any of AD within 4 weeks (or 5 half-lives, whichever is longer) prior to screening;
20. Has received phototherapy (narrow-band ultraviolet B [NBUVB], ultraviolet B [UVB], ultraviolet A1 [UVA1], psoralen + ultraviolet A [PUVA]), tanning beds, or any other light-emitting device within 4 weeks prior to screening;
21. Those who have used any strong inhibitor or inducer of any CYP3A4 enzyme within 4 weeks prior to screening (strong inhibitors include clarithromycin, itraconazole, ketoconazole, ritonavir, and strong inducers include rifampin and phenytoin);
22. Received topical drug therapies known or likely to affect AD within 2 weeks (or 5 half-lives, whichever is longer) before screening, including but not limited to topical TCS, TCI, topical PDE-4 inhibitors, topical JAK inhibitors, etc.;
23. Consumption of excessive amounts of tea, coffee, and/or caffeinated beverages (more than 8 cups, 1 cup = 250 mL) per day for 2 weeks prior to screening;
24. Intake of food or beverages (e.g. tea, coffee, cola, energy drinks or chocolate) containing grapefruit and/or grapefruit, caffeine, and/or xanthine from 48 h before dosing until leaving the ward;
25. Other conditions or treatments that, as assessed by the investigator, may affect the results of the study, interfere with the participation of participants in the trial, etc.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-09-12 (Actual); Primary Completion 2026-09-09 (Estimated); Study Completion 2026-09-09 (Estimated)

PRIMARY OUTCOMES:
Adverse Events assessed by CTCAE V5.0 | Part1:Day20；Part2:Day36
  The latest version of the Regulatory Activity Medical Dictionary (MedDRA) was used to encode AE terms used by investigators in eCRF. All adverse events (TEAE) that occurred during treatment were analyzed. TEAE will be summarized by dose grouping by systematic organ classification, preferred terminology and CTCAE classification, and relationship to investigational drug products.
Vital signs | Part1: Day-7~Day-1，Day-1，Day1~Day13，Day20；Part2: Day-14~Day-2，Day-1，Day1，Day2，Day7, Day8，Day15, Day29，Day36
  Summary changes in heart rate, blood pressure (systolic and diastolic), body temperature (frontal temperature), and respiratory rate, as well as relative baseline levels, were descriptively summarized at each planned time point.
  The changes of clinical significance before and after physical examination and treatment will be described.
12-lead electrocardiogram | Part1: Day-7~Day-1，Day-1，Day1~Day13，Day20；Part2: Day-14~Day-2，Day-1，Day1，Day2，Day7, Day8，Day15, Day29，Day36
  Including PR interval, QRS interval, QT interval and QTc interval. To provide a descriptive summary of changes in ECG parameters relative to baseline by visit, and to provide a summary of changes in clinical significance of ECG parameters before and after treatment.
Laboratory examination | Part1: Day-7~Day-1，Day13，Day20；Part2: Day-14~Day-2，Day-1， Day8，Day15, Day29，Day36
  The data of laboratory tests were summarized according to the type of laboratory tests, and the changes of laboratory test values at baseline and post-treatment planned time points and relative baseline levels were descriptively summarized, and the changes in clinical significance before and after treatment were provided.
Skin tolerance assessment | Part1: Day1~Day20；Part2: Day1~Day36
  Descriptive summary of skin tolerances. Skin tolerance was assessed based on local irritant reactions (e.g. rash, redness, pain, etc.) to the participant's skin at the time points specified in the SoA. If the skin tolerance problems described above occur after a participant receives the study treatment and are assessed by the investigator as abnormal and clinically significant, an AE should be recorded and adverse event generics performed.Language Standards (CTCAE) v5.0 assessment criteria were used to assess their severity.
Physical examination | Part1: Day-7~Day-1，Day-1，Day1，Day4~Day9，Day10，Day13，Day20；Part2: Day-14~Day-2，Day-1，Day1，Day7, Day8，Day15, Day29，Day36
  This includes general examination, examination of the skin and mucous membranes, lymph nodes, head, neck, chest, abdomen, spine, and limbs, or other areas as needed.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No